CLINICAL TRIAL: NCT00801983
Title: The Effect of Alternative Keyboards on Discomfort and Typing Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Baker, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 08030467; R01OH008961 (NIH)
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Subject receives typical keyboard first for 6 months and alternative keyboard second for 6 months
  Interventions: Device: Alternative Keyboard
- B (Experimental): Subject receives alternative keyboard first for 6 months and typical keyboard second for 6 months
  Interventions: Device: Alternative Keyboard

INTERVENTIONS:
Device: Alternative Keyboard — Subjects use either a typical or alternative keyboard
  Other Names: Microsoft Natural Ergonomic

SUMMARY:
Awkward postures during computer keyboard use have been hypothesized to be one cause of musculoskeletal pain/discomfort as well as musculoskeletal disorders of the upper extremity (MSD-UE). Alternative computer keyboards purport to reduce musculoskeletal pain/discomfort and have been shown to change aspects of keyboard users' kinematics under laboratory conditions. However, research that has examined the effectiveness of alternative keyboards in reducing musculoskeletal pain/discomfort in the workplace is equivocal, and no study has examined the association between postures and musculoskeletal pain. The Aims of this 3-year prospective double cross-over trial are: 1) To examine the effectiveness of an alternative keyboard in reducing reports of pain over 6-months; 2) To examine the neutrality and stability of postures during keyboard use; and 3) To identify which postures are associated with lower levels of musculoskeletal pain. Seventy-five computer users will be randomly assigned to one of two keyboard use orders: Group 1 - AB (standard keyboard, alternative keyboard); Group 2 - BA (alternative keyboard, standard keyboard). All subjects will use their assigned keyboards for 6-months before switching to the next keyboard. Every week, subjects will report their musculoskeletal pain levels. Just prior to and just after each 6-month intervention subjects' kinematics performances on the keyboards will be recorded at the worksite using the Keyboard - Personal Computing Style (K-PeCS) instrument and in a laboratory setting using 3-dimensional motion capture technology.

Aim 1: To examine the effectiveness of an alternative keyboard in reducing pain over 6-months.

Hypothesis 1 (H-1) - At six months subjects using an alternative keyboard will have significantly lower musculoskeletal pain levels than when using a standard keyboard.

Aim 2: To examine the neutrality and stability of postures during keyboard use.

Hypothesis 3 (H-2) - Subjects using an alternative keyboard will have significantly more neutral postures than when using a standard keyboard at baseline and at 6 months Hypothesis 3 (H-3) - Subjects 6-months keyboarding postures will remain equivalent to the keyboarding postures documented at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Use a computer at least 20 hrs per week
* Aged 18-65
* Experiencing some pain during computer use

Exclusion Criteria:

* Currently use an alternative keyboard
* Serious trauma injury to the upper extremity
* Rheumatic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Typical/Alternative): Subject receives typical keyboard for 5-6 months first and alternative keyboard second for 5-6 months (total 12 months in study
- Group B (Alternative/Typical): Subject receives alternate keyboard for 5-6 months first and typical keyboard second for 5-6 months (total 12 months in study
Period: Period 1
Arm/Group | Group A (Typical/Alternative) | Group B (Alternative/Typical)
Started | 44 | 41
Completed | 40 | 33
Not Completed | 4 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 8
Period: Period 2
Arm/Group | Group A (Typical/Alternative) | Group B (Alternative/Typical)
Started | 40 | 33
Completed | 38 | 32
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: GEE analyses allows a subjects inclusion even if they did not complete the full trial. Although we had a total of 15 subjects not complete the full trial we had sufficient data on 77 subjects to complete the GEE statistical analyses. With the crossover design we compared 77 subjects using the standard keyboard to 77 subjects using the alternative
Groups:
- Group A: Subject receives typical keyboard first (0-6 months) and alternative keyboard second (7-12 months). In this crossover design all subjects received both standard and alternative keyboard, each group just received the keyboards in a different order
- Group B: Subject receives alternative keyboard first (0-6 months) and typical keyboard second (7-12 months). In this crossover design all subjects received both standard and alternative keyboard, each group just received the keyboards in a different order
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 40 | 37 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.9) | 45.6 (11.9) | 44.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 36 | 31 | 67
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 37 | 77
Avg Computer Use [Mean (Standard Deviation); unit: hrs/day] | 6.3 (1.1) | 6.1 (1.5) | 6.2 (1.3)
Typing Speed [Number; unit: participants]
  Slow | 7 | 3 | 10
  Moderately Fast | 16 | 14 | 30
  Fast | 11 | 12 | 23
  Don't know | 6 | 8 | 14
Baseline Discomfort [Number; unit: participants]
  Neck (Yes) | 36 | 36 | 72
  Back (Yes) | 33 | 33 | 66
  Right arm hand (Yes) | 33 | 36 | 69
  Left Arm hand (Yes) | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Musculoskeletal Discomfort
Description: Discomfort Survey (WDS) was used to assess symptoms and activity limitations. Participants reported on their work schedule, medication used for pain control, and discomfort in their neck/shoulder, back, and bilateral lower arms (elbows, forearms, wrists, and hands) using an 11-point numerical rating scale (0 = no discomfort/no limitations; 10 = unbearable discomfort/major limitations).
  We had to dichotomize the data during analysis due to severe skew towards not discomfort (0). Thus the final outcome was discomfort -yes or no
Time Frame: 6 months and 12 months
Measure: Number; unit: percentage of subjects with MSD
Groups:
- Typical Keyboard: MSD reported when a subject was typing on a typical keyboard (regardless of order)
- Alternative Keyboard: MSD reported when a subject was typing on an alternative keyboard (regardless of order)
Arm/Group | Typical Keyboard | Alternative Keyboard
Number analyzed (Participants) | 77 | 77
percentage of subjects with MSD | 20 | 20
Statistical Analysis 1: Comparison: Typical Keyboard vs Alternative Keyboard; Subjects were compared across keyboard types - The percentage of subjects with MSD when using the alternative keyboard were compared to the % of subjects with MSD when they were using the typical keyboard; Test type: Superiority or Other; p > .05, GEE

ADVERSE EVENTS:
Arm/Group | Typical Keyboard | Alternative Keyboard
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No